CLINICAL TRIAL: NCT06619054
Title: An Open-label, Single-dose Study for the Evaluation of the Effect of Hepatic Impairment on the Pharmacokinetics and Safety of KP-001
Brief Title: A Study to Evaluate the Effect of Hepatic Impairment on the Pharmacokinetics of KP-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kaken Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KP-001-105
Record Dates: First submitted 2024-09-12; First posted 2024-10-01 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Healthy Adults; Hepatic Impairment

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort1 (Normal) (Experimental): Child-Pugh Score: N/A
  Interventions: Drug: KP-001
- Cohort2 (Mild Impairment) (Experimental): Child-Pugh Score: A (5 to 6 points)
  Interventions: Drug: KP-001
- Cohort3 (Moderate Impairment) (Experimental): Child-Pugh Score: B (7 to 9 points)
  Interventions: Drug: KP-001
- Cohort4 (Severe Impairment) (Experimental): Child-Pugh Score: C (10 to 15 points)
  Interventions: Drug: KP-001

INTERVENTIONS:
Drug: KP-001 — Oral single dose 50mg.

SUMMARY:
This is a phase 1, open-label, non-randomized, parallel-group, single-dose study to assess the effect of hepatic impairment (assessed by the criteria of the Child-Pugh scale) on the pharmacokinetics (PK) and safety of KP-001 in adult male and non-childbearing potential female participants aged ≥20 years old.

The purpose of this study is to evaluate the effect of hepatic impairment on the PK and safety of KP-001. The study will also assess the effect of hepatic impairment on other PK parameters after single dose administration of KP-001.

The study will comprise 3 parts, and the study period for each part will consist of the following:

* Screening period: Up to 28 days before the administration of study intervention
* Treatment Period: Participants will be residential at the Clinical Unit from the day before the administration of the single dose of KP-001 (Day -1) until Day 3 (Discharge)
* Follow-up Visit: 7 days after discharge from the Clinical Unit (ie, Day 10) Participants will be enrolled into 4 cohorts according to the hepatic function status as summarized below. The study includes a control group of healthy participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

・All Participants (Cohorts 1 to 4)

1. Participant is male or female and aged ≥20 years old at the time of signing the informed consent.
2. Participant has body weight ≥40.0 kg and body mass index between 18.0 and 42.0 kg/m2 at screening.
3. Female participant is a woman of non-childbearing potential who:

   1. Is postmenopausal with amenorrhea for at least 1 year prior to screening and with FSH of 40 IU/L or higher.

      OR
   2. Has undergone one of the following:

      * bilateral tubal ligation or bilateral salpingectomy
      * hysterectomy
      * bilateral oophorectomy
4. Male participant who is sexually active with female partner(s) of childbearing potential must agree to use both a condom and spermicide from the day of the administration of KP-001 until 91 days after the administration of KP-001.
5. Male participant must agree to not donate sperm from the day of the administration of KP-001 until 91 days after the administration of KP-001.
6. Participant is capable of giving signed informed consent as described in Appendix 1, Section 10.1.3 which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

   ・Healthy Participants with Normal Hepatic Function (Cohort 1)
7. Participant is of a gender matched to his/her matched participant enrolled in Cohort 3.
8. Participant is of an age that is within ±10 years to his/her matched participant enrolled in Cohort 3.
9. Participant has a body mass index within ±20% to his/her matched participant enrolled in Cohort 3.
10. Participant is medically healthy with no clinically significant abnormal screening results (e.g., medical history, physical examination, laboratory profiles, vital signs, or ECGs), in the opinion of the Investigator or designee.

    If screening and/or admission results are abnormal, they may be repeated once at screening and/or once at admission to confirm the participant's eligibility.
11. Participant whose AST and ALT at screening and admission meet the following: ALT and AST &amp;amp;amp;lt; 2 ULN.
12. Participant has negative results for hepatitis B, hepatitis C, and HIV antibody screens.
13. Non-smoker and no use of other tobacco- or nicotine-containing products, as documented by history (no tobacco or nicotine use within 6 months prior to Screening) during the study.

    ・Participants with Hepatic Impairment (Cohorts 2 to 4)
14. Participant whose Child-Pugh classification at screening and admission laboratory tests applies to any of the following:

    * Cohort 2: Child-Pugh Grade A (score 5-6)
    * Cohort 3: Child-Pugh Grade B (score 7-9)
    * Cohort 4: Child-Pugh Grade C (score 10-15)
15. Participant considered by the Investigator to be clinically stable with respect to underlying hepatic impairment, based on medical evaluation that includes medical and surgical history, as well as a complete physical examination including seated vital signs, 12-lead ECG, and laboratory test results.
16. Participant whose laboratory abnormalities are judged by the investigator to be clinically acceptable.
17. Participant has no clinical exacerbation of hepatic disease within 30 days prior to study intervention administration.
18. Participant with negative hepatitis B surface antigen (HBsAg) at screening.
19. Non-smoker and no use of other tobacco or nicotine-containing products during the study.

Exclusion Criteria:

・All Participants (Cohorts 1 to 4)

1. Participant has a history or presence of hypersensitivity or idiosyncratic reaction to any components of the KP-001 formulation or any components of formulation used as study intervention during the study.
2. Participant has a complication of drug allergies or history of drug allergies, or psychiatric disorder as determined by the Investigator or designee.
3. Participant used any investigational drug in the last 30 days or 5 half-lives (if known), whichever is longer, prior to Day -1 of Treatment Period.
4. Female participant has a positive pregnancy test or is lactating.
5. Participant has positive urine drug or urine alcohol and positive cotinine test results at screening or Day -1 of Treatment Period.
6. Participant who cannot administer drugs orally.
7. Participant is unable or unwilling to undergo multiple venipunctures.
8. Participant underwent blood donation or transfusion within 56 days prior to Day -1 of Treatment Period.
9. Participant has consumed alcohol- or caffeine-containing foods and beverages within 72 hours prior to Day -1 of Treatment Period and does not agree to refrain from consuming during the entire study, unless deemed acceptable by the Investigator.
10. Participant has consumed grapefruit-containing foods and beverages within 7 days prior to Day -1 of Treatment Period and does not agree to refrain from consuming during the entire study.
11. Participant has consumed St. John's wort-containing foods and beverages within 14 days prior to Day -1 of Treatment Period and does not agree to refrain from consuming during the entire study.
12. Participated in strenuous exercise from 48 hours prior to Check-in (Day -1) or during the study through the final end of study assessment.
13. Participant is legally, mentally or physically incapacitated or, in the opinion of the Investigator, has significant mental or emotional problems, including psychiatric illness (e.g., depression and/or anxiety) at the time of the Screening Visit, or that could reasonably be expected to develop during the conduct of the study.
14. Participant had any laboratory abnormality that, in the judgment of the Investigator, would put the participant at unacceptable risk for participation in the study or may interfere with the assessments included in the study.
15. Participant has abnormal findings on the screening ECG deemed clinically significant by the Investigator or qualified designee.
16. Participant is an employee of the Sponsor or any CRO involved in the study, the Investigator, or an immediate family member (partner, offspring, parents, siblings, or sibling's offspring) of an employee involved in the study.
17. Any other reason that would render the participant unsuitable for study enrollment at the discretion of the Investigator.
18. A participant who has received proton pump inhibitors (PPIs), histamine type-2 (H2)-receptor antagonists, or antacids during the 5-day period immediately preceding and including the admission day (or for 5 half-lives of the medication whichever is longer), or plan to receive any of these medications during treatment period (ie, until Day 3 [Discharge]).

    ・Healthy Participants with Normal Hepatic Function (Cohort 1)
19. Participant has a significant history or clinical manifestation of any metabolic, allergic, dermatologic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder as determined by the Investigator or designee.
20. Participant has a history of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
21. Participant had any major illness within 30 days before the Screening Visit.
22. Participant had any major surgical procedure within 30 days prior to Day -1 of Treatment Period or any planned surgery during study period.
23. Participant has a history or presence of liver disease or cholecystectomy within one year prior to screening.
24. Participant has a disorder or any condition that would interfere with the absorption, distribution, metabolism, or excretion of drugs.
25. Participant used any prescription or non-prescription medications (including vitamins, recreational drugs, and dietary or herbal supplements) within 14 days or 5 half-lives (whichever is longer) prior to Day -1 of Treatment Period and until completion of the Followup Visit unless, in the opinion of the Investigator, may be treatment for an AE or will not interfere with the interpretation of safety.

    ・Participants with Hepatic Impairment (Cohorts 2 to 4)
26. Participant with any concomitant disease or condition considered clinically significant that, in the opinion of the investigator, may interfere with the investigational product, pose an unacceptable risk to the participant, or significantly increase the risk to the integrity or utility of the trial data (including treatment of such conditions).
27. Participant with acute or chronic conditions other than liver (including, but not limited to, poorly controlled diabetes and grade 3 or higher encephalopathy) that, in the opinion of the investigator, would limit the participant&amp;amp;amp;#39;s ability to complete the study and/or participate in this study.
28. Participant with acute exacerbation of liver dysfunction or unstable liver function as determined by the investigator by Day 1 from screening.
29. Participant who is positive for HBsAg, hepatitis C or HIV at screening. Participants with hepatitis C will also be accepted if, in the investigator&amp;amp;amp;#39;s judgement, they are clinically stable and not receiving active treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
PK parameters of KP-001 in plasma: Cmax | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
  To evaluate the effect of hepatic impairment on the PK and safety of KP-001
PK parameters of KP-001 in plasma:AUC0-inf | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
  To evaluate the effect of hepatic impairment on the PK and safety of KP-001

SECONDARY OUTCOMES:
PK parameters of KP-001 in plasma: AUC0-last | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
  To assess the effect of hepatic impairment on other PK parameters after single dose administration of KP-001
PK parameters of KP-001 in plasma: t1/2 | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
  To assess the effect of hepatic impairment on other PK parameters after single dose administration of KP-001
PK parameters of KP-001 in plasma: λz | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
  To assess the effect of hepatic impairment on other PK parameters after single dose administration of KP-001
PK parameters of KP-001 in plasma: CL/F | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
  To assess the effect of hepatic impairment on other PK parameters after single dose administration of KP-001
PK parameters of KP-001 in plasma: Vz/F | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
  To assess the effect of hepatic impairment on other PK parameters after single dose administration of KP-001
PK parameters of KP-001 in plasma: Tmax | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
  To assess the effect of hepatic impairment on other PK parameters after single dose administration of KP-001

CONTACTS AND LOCATIONS:
Locations (1):
- Sites contracted by Parexel, San Antonio, Texas, United States